CLINICAL TRIAL: NCT07260227
Title: Influence of a PSychological Intensive Support Program for Lung Cancer Patients ON Post-operative Outcomes: a Prospective Clinical Trial (IPSILON Trial).
Brief Title: Influence of a PSychological Intensive Support Program for Lung Cancer Patients ON Post-operative Outcomes.
Acronym: IPSILON
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8086
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: NSCLC; Anxiety Postoperative; Depression
MeSH Terms: conditions — Depression | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Group (Experimental): patients who resulted anxious at psychological tests who accepted the intensive psychological support
  Interventions: Other: HADS (Hospital Anxiety and Depression Scale)
- Pathological Control Group (Active Comparator): patients who resulted anxious at psychological tests who refused the intensive psychological support
  Interventions: Other: HADS (Hospital Anxiety and Depression Scale)
- Healthy Control Group (Active Comparator): patients who resulted not anxious at psychological tests
  Interventions: Other: HADS (Hospital Anxiety and Depression Scale)

INTERVENTIONS:
Other: HADS (Hospital Anxiety and Depression Scale) — The psychological treatment, for those patients who accepted the enrollment, consists of a weekly 45-minute psychological session for 4 weeks before the recovery in the thoracic department for lung resection. Measurement of psychological test will be collected at the first visit (T0), the day before surgery (T1) and 30 day after surgery (T3); VAS and ISI measurements were collected at T1, the day after surgery (T2) and 30 day after surgery (T3).
  Other Names: psychological evaluation

SUMMARY:
Anxiety is common among patients diagnosed with lung cancer, affecting 50-60% of cases, and over 30% report moderate to severe psychological distress. This distress includes symptoms such as depression, anxiety and social withdrawal. The waiting period before lung resection often heightens emotional tension due to fears about reduced respiratory function and postoperative dyspnea. Persistent anxiety may continue during follow-up because of the risk of recurrence and the potential need for adjuvant therapy. Previous studies have shown that high perioperative anxiety is associated with longer hospitalization, increased complications, particularly delirium and cardiac arrhythmias, and poorer adherence to treatment.

This study aims to assess whether a brief, intensive preoperative psychological intervention reduces anxiety levels in lung cancer patients, measured using the Hospital Anxiety and Depression Scale (HADS). Scores of 0-7 indicate normal levels, ≥ 8 probable anxiety or depression. Additional tools include the Visual Analogue Scale (VAS) for pain (0 = no pain, 10 = worst pain imaginable) and the Insomnia Severity Index (ISI) (0-7 no insomnia, 8-14 subthreshold, 15-21 moderate, 22-28 severe). At hospital discharge, patients were invited to complete a questionnaire about satisfaction. Measurement of psychological test will be collected at the first visit (T0), the day before surgery (T1) and 30 day after surgery (T3); VAS and ISI measurements were collected at T1, the day after surgery (T2) and 30 day after surgery (T3).

Patients are divided into three groups: an intervention group receiving four weekly 45-minute psychological sessions, a pathological control group refusing support, and a healthy control group without anxiety. Primary outcomes are changes in HADS scores between T0 and T1; secondary outcomes include complications, pain, insomnia, length of stay, and patient satisfaction. The study is a twelve-month prospective controlled trial with an estimated 46 patients per group

ELIGIBILITY:
Inclusion Criteria:

* age more than 18
* candidate to thoracic resection for lung cancer with radical intent
* consent to participate in the research study.

Exclusion Criteria:

* synchronous cancer requiring chemo or radiotherapy
* history of chronic pain, vulnerable patients (e.g., minors and/or incapacitated subjects)
* patients with severe psychiatric conditions (psychosis and/or personality disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale HADS | 1 day
  The primary endpoint is the reduction in anxiety and depression as measured by the subscales of the Hospital Anxiety and Depression Scale (HADS) between T0 and T1 among the study groups.

SECONDARY OUTCOMES:
evaluation of the incidence of complications | 1 month
  Secondary endpoints are to evaluate the incidence of complications (in terms of delirium, cardiac complications), perception of pain, insomnia and length of stay in the study group compared to the two control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Teresa Congedo, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS